CLINICAL TRIAL: NCT03455621
Title: Effect of the Amount of Fluoride Toothpaste on Fluoride Availability in the Oral Fluids in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Livia Maria Andaló Tenuta, Associate Professor, University of Campinas, Brazil
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: FOPBioq007
Record Dates: First submitted 2018-02-21; First posted 2018-03-06 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-02

CONDITIONS: Dental Caries
Keywords: dental caries; fluoride; toothpaste; dentifrice
MeSH Terms: conditions — Dental Caries | interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Pea-size amount of non-F dentifrice (Placebo Comparator): Non-fluoride dentifrice (0 ppm F); to be used twice/day. Amount to be used: 0.3 g (pea-size amount)
  Interventions: Procedure: Toothbrushing
- 0.025 g of 1,100 ppm F dentifrice (Experimental): Fluoride dentifrice (1,100 ppm F, as NaF); to be used twice/day. Amount to be used: 0.025 g
  Interventions: Procedure: Toothbrushing
- 0.05 g of 1,100 ppm F dentifrice (Experimental): Fluoride dentifrice (1,100 ppm F, as NaF); to be used twice/day. Amount to be used: 0.05 g
  Interventions: Procedure: Toothbrushing
- 0.1 g of 1,100 ppm F dentifrice (Experimental): Fluoride dentifrice (1,100 ppm F, as NaF); to be used twice/day. Amount to be used: 0.1 g
  Interventions: Procedure: Toothbrushing
- Pea-size amount of 1,100 ppm F dentifrice (Active Comparator): Fluoride dentifrice (1,100 ppm F, as NaF); to be used twice/day. Amount to be used: 0.3 g (pea-size amount)
  Interventions: Procedure: Toothbrushing

INTERVENTIONS:
Procedure: Toothbrushing — Toothbrushing with different amounts of fluoride toothpaste (or a non-fluoride toothpaste as a control)

SUMMARY:
The aim of the study is to determine the fluoride availability in saliva and dental biofilm after the use of increasing amounts of fluoride toothpaste. Using a crossover and blind design, 15 children (18-42 months old) had their teeth brushed with increasing amounts of fluoride toothpaste. Fluoride concentration in saliva and dental biofilm was determined up to 30 min after brushing.

DETAILED DESCRIPTION:
The aim of the study is to determine the fluoride availability in saliva and dental biofilm after the use of increasing amounts of fluoride toothpaste. Children from 18 to 42 months from a community daycare participated. The study had a crossover and blind design. The amounts of toothpastes tested were: 1. A pea-size amount (0.3 g) of a non-F toothpaste; 2. 0.025 g of a F toothpaste (1,100 ppm F, as NaF); 3. 0.05 g of the same F toothpaste; 4. 0.1 g of the same F toothpaste; or 5. 0.3 g (pea-size) of the same F toothpaste. Children were to brush their teeth with the designated amount of toothpaste twice/day from Monday to Friday. In order to allow biofilm accumulation, caregivers were instructed to brush only the occlusal surfaces of primary molars. On Friday morning, at least one hour after breakfast, saliva and one biofilm sample from the right or left hemiarch were collected and analyzed for fluoride concentration. Then, brushing with the respective amount of toothpaste was performed, and saliva was collected 5, 15 and 30 min later. The biofilm from the other side of the mouth was collected after 30 min. Fluoride concentration in saliva and biofilm samples was determined with an ion-specific electrode.

ELIGIBILITY:
Inclusion Criteria:

* All children with an informed consent signed by the parents/guardians

Exclusion Criteria:

* Children with at least on active caries lesion

Ages: 18 Months to 42 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2010-03-01 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2011-06-30 (Actual)

PRIMARY OUTCOMES:
Fluoride concentration in saliva before brushing | Before brushing (baseline)
Fluoride concentration in saliva 5 min after brushing | 5 minutes after brushing
Fluoride concentration in saliva 15 min after brushing | 15 min after brushing
Fluoride concentration in saliva 30 min after brushing | 30 min after brushing
Fluoride concentration in dental biofilm (fluid fraction) before brushing | Before brushing (baseline)
Fluoride concentration in dental biofilm (fluid fraction) 30 min after brushing | 30 min after brushing
Fluoride concentration in dental biofilm (solid fraction) before brushing | Before brushing (baseline)
Fluoride concentration in dental biofilm (solid fraction) 30 min after brushing | 30 min after brushing

IPD SHARING:
Plan to Share IPD: No